CLINICAL TRIAL: NCT06459869
Title: A Multicentre, Open-label, Non-randomized, Phase 1b Trial of NG-350A, a Tumour-selective Anti-CD40-expressing Adenoviral Vector, in Combination With Chemoradiotherapy in Locally Advanced Rectal Cancer (FORTRESS)
Brief Title: NG-350A Plus Chemoradiotherapy for Locally Advanced Rectal Cancer
Acronym: FORTRESS
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Akamis Bio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NG-350A-03; https://www.FortressStudy.org (Other: Akamis Bio)
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-08

CONDITIONS: Locally Advanced Rectal Cancer (LARC)
Keywords: Treatment naive; Oligometastatic
MeSH Terms: interventions — Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NG-350A plus CRT during a 12-week active study treatment period (Experimental)
  Interventions: Drug: NG-350A IV administration; Drug: Capecitabine oral administration; Radiation: Radiotherapy

INTERVENTIONS:
Drug: NG-350A IV administration — a tumour-selective anti-CD40-expressing adenoviral vector
Drug: Capecitabine oral administration — chemotherapy
Radiation: Radiotherapy — long-course intensity-modulated radiotherapy

SUMMARY:
The FORTRESS trial (NG-350A-03) is an open-label, single-arm, and multicentre trial of NG-350A in combination with chemoradiotherapy (CRT) in adult patients with locally advanced rectal cancer (LARC) and at least one risk factor for local or distant recurrence.

ELIGIBILITY:
Selected Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the rectum.
* Locally advanced disease (clinical stage II-III based on pelvic MRI) selected by a multidisciplinary team for treatment with neoadjuvant CRT (which may be followed by CNCT to comprise planned TNT). Patients with oligometastatic disease are permitted provided that the site-specific multidisciplinary team deems them suitable for radical treatment/chemoradiation.
* Confirmed microsatellite stable (MSS)/proficient mismatch repair (pMMR) status.
* Provide written informed consent to participate.
* ECOG Performance Status 0 or 1.
* Must not be pregnant or breastfeeding.
* Patients who are sexually active (with either sex) must agree to comply with contraceptive requirements.
* Adequate lung reserve, renal function, hepatic function, and bone marrow/hematological function assessed ≤ 10 days prior to first dose.

Selected Exclusion Criteria:

* Recurrent rectal cancer.
* Distant metastatic disease not amenable to radical treatment/chemoradiation.
* Other prior malignancy active within the previous 3 years, except for local or organ confined early-stage cancer that has been definitively treated with curative intent, does not require ongoing treatment, has no evidence of residual disease, and has a negligible risk of recurrence and is therefore unlikely to interfere with the primary and secondary endpoints of the trial, including response rate and safety.
* Splenectomy (patients with prior partial resection remain eligible if the Investigator considers splenic function to not be significantly compromised).
* Active autoimmune disease that has required systemic therapy in the past 2 years, immunocompromised status in the opinion of the Investigator, or current treatment with systemic immunosuppressive therapy (daily prednisone equivalent for chronic system replacement not to exceed 10mg per day).
* Infectious or inflammatory bowel disease in the 3 months before the first dose of study treatment.
* Any clinically significant cardiovascular, peripheral vascular, cerebrovascular, or thromboembolic event in the last 1 month before the first dose of study treatment.
* Major surgery in the 14 days before the first dose of study treatment or any surgical wounds that are not fully healed and free of infection or dehiscence.
* Any prior surgery for rectal cancer or pelvic radiotherapy.
* Any other anti-cancer or experimental therapy within the previous 12 months or that is planned during the active study treatment period.
* Treatment with any other enadenotucirev-based virus (parent virus or transgene-modified variants), or anti-CD40 antibody at any time.
* History of prior Grade 3-4 acute kidney injury or other clinically significant renal impairment.
* Any ongoing Common Terminology Criteria for Adverse Events (CTCAE) Grade ≥2 coagulation abnormality/coagulopathy.

URL:

https://www.FortressStudy.org

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving a clinical complete response (cCR) | 12 weeks after initiating NG-350A in combination with chemoradiotherapy (CRT)

SECONDARY OUTCOMES:
Incidence and severity of adverse events graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0 | 1-3 years
Clinical response (CR) outcome | 12, 18, and 36 weeks after initiating NG-350A plus chemoradiotherapy (CRT)
MRI-based tumor regression grade (mrTRG) | 12, 18, and 36 weeks after initiating NG-350A plus chemoradiotherapy (CRT)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (4):
  - AdventHealth Orlando, Orlando, Florida
  - Washington University School of Medicine, St Louis, Missouri
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- United Kingdom (2):
  - University College London NHS FT, London
  - The Royal Marsden NHS Foundation Trust, Sutton

REFERENCES:
- [Derived] Naing A, Khalil D, Rosen O, Camidge DR, Lillie T, Ji RR, Stacey A, Thomas M, Rosen L. First-in-human clinical outcomes with NG-350A, an anti-CD40 expressing tumor-selective vector designed to remodel immunosuppressive tumor microenvironments. J Immunother Cancer. 2024 Oct 15;12(10):e010016. doi: 10.1136/jitc-2024-010016. PMID 39414325
- See also: Fortress Study Information — https://www.FortressStudy.org